CLINICAL TRIAL: NCT04764929
Title: Helmet CPAP for Infants and Pediatric Patients With Acute Respiratory Distress
Brief Title: Pediatric Helmet CPAP Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigators left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT5640
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Bronchiolitis, Viral; Pneumonia, Viral; Pneumonia, Bacterial
MeSH Terms: conditions — Bronchiolitis, Viral; Pneumonia, Viral; Pneumonia, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Helmet CPAP (Experimental): Patients in the Pediatric Intensive Care Unit (PICU) already receiving CPAP through a facemask or nasal prongs or mask for at least four hours but no more than 48 hours will be transitioned to the Vyatil nonpowered oxygen tent system (Rochester, NY) by trained respiratory therapists per the manufacture's instructions: patient's neck circumference will be measured with a soft tape measure to ensure appropriate sizing. The helmet will be connected to at least 30 liters per minute of high flow medical air with an oxygen blender. The expiratory limb will be attached to the positive end expiratory pressure (PEEP) valve (initially set at 5 centimeters of water pressure) connected to a high-efficiency particulate air (HEPA) filter to prevent any viral particles from being released into the environment. A disposable manometer will be used to measure the pressure within the helmet. Once the flow to the helmet interface is on, the helmet will be sealed and secured with the system's arm straps.
  Interventions: Device: Helmet CPAP

INTERVENTIONS:
Device: Helmet CPAP — Vyatil nonpowered oxygen tent system

SUMMARY:
This a research study to find out whether giving Continuous Positive Airway Pressure (CPAP) through a Helmet is the same or better than giving CPAP through a Facemask, Nasal Mask, or Nasal Prongs. CPAP can help kids with lung infections breathe easier. The machine delivers pressurized air, which may help people with lung infections breathe more easily. Doctors routinely use a Facemask, Nasal Mask or Nasal Prongs to give CPAP for kids with lung infections, but the researchers want to know whether using Helmet CPAP is the same or better.

DETAILED DESCRIPTION:
Prior clinical trials have demonstrated efficacy of Helmet CPAP in adults with acute respiratory distress syndrome, superior tolerance and improved respiratory scores compared to nasal/facial CPAP in infants, and no major safety concerns were identified with the use of helmet CPAP. This is a prospective pilot study to (1) determine if infants and pediatric patients requiring CPAP in the PICU will tolerate helmet CPAP for at least four hours, and (2) measure changes in the respiratory rate, oxygen saturation, heart rate and blood pressure over four hours. If helmet CPAP is found to be well tolerated in this small cohort, a larger study comparing it directly to other CPAP interfaces will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* One month to 5 years of age (inclusive) admitted to the PICU with community acquired pneumonia or bronchiolitis, having been stable on nasal or facemask CPAP for at least four hours but less than 48 hours, and parental informed consent.

Exclusion Criteria:

* Age less than 1 month or greater than 5 years
* Positive for COVID-19
* Need for invasive mechanical ventilation or higher levels of non-invasive ventilation such as bi-level positive airway pressure (BPAP)
* Unresponsiveness (GCS 8 or less)
* Hypotension as defined as a systolic blood pressure less than 5th percentile for age
* Existing head or neck trauma, known or suspected air leak syndrome (pneumothorax, pneumomediastinum, subcutaneous emphysema), known or suspected increased intracranial pressure
* Non-English speaking parent

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Helmet CPAP
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Helmet CPAP
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Admission Diagnosis [Count of Participants; unit: Participants]
  Viral Bronchiolitis | 3
  Viral Pneumonia | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Tolerated CPAP Helmet for at Least Four Hours
Description: Tolerance is defined as the successful application and maintenance of helmet CPAP without any unplanned, prolonged (>5 minutes) removals or disruptions.
Time Frame: Four hours
Measure: Count of Participants; unit: Participants
Arm/Group | Helmet CPAP
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Respiratory Rate
Description: Respiratory rate will be measured in breaths per minute every hour for four hours.
Time Frame: 4 hours
Population: Data was not collected thus cannot be analyzed or reported.
Arm/Group | Helmet CPAP
Number analyzed (Participants) | 0

3. Secondary Outcome: Heart Rate
Description: Heart rate will be measured in beats per minute every hour for 4 hours.
Time Frame: 4 hours
Population: Data was not collected thus cannot be analyzed or reported.
Arm/Group | Helmet CPAP
Number analyzed (Participants) | 0

4. Secondary Outcome: Oxygen Saturation
Description: Pulse oxygen saturation will be measured as a percent every hour for 4 hours.
Time Frame: 4 hours
Population: Data was not collected thus cannot be analyzed or reported.
Arm/Group | Helmet CPAP
Number analyzed (Participants) | 0

5. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure will be measured in millimeters of mercury every hour for 4 hours.
Time Frame: 4 hours
Population: Data was not collected thus cannot be analyzed or reported.
Arm/Group | Helmet CPAP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 hours
Arm/Group | Helmet CPAP
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04764929/Prot_001.pdf